CLINICAL TRIAL: NCT04646018
Title: The Effect of Lumbopelvic Non-Thrust Spinal Manipulation on Muscle Thickness of the Sacral Multifidi, Lumbar Motion, and Self-Reported Pain
Brief Title: The Effect of Lumbopelvic Non-Thrust Spinal Manipulation on Individuals With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alvernia University (Other)
Responsible Party: Principal Investigator, Christopher H. Wise, Physical Therapy Department Chair, Professor of Physical Therapy, Alvernia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AlverniaU
Record Dates: First submitted 2020-11-05; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar Manipulation Group (Experimental): Group that receives experimental lumbar non-thrust manipulation
  Interventions: Other: Lumbar Spine Manipulation
- Sham Manipulation Group (Sham Comparator): Group that receives sham lumbar non-thrust manipulation
  Interventions: Other: Sham Manipulation

INTERVENTIONS:
Other: Lumbar Spine Manipulation — Lumbar non-thrust manipulation is a passive movement that is performed with a rhythm and a grade in a manner in which the patient is able to prevent the technique from being performed.
  Arms: Lumbar Manipulation Group
Other: Sham Manipulation — Lumbar non-thrust manipulation without force applied
  Arms: Sham Manipulation Group

SUMMARY:
The purpose of this experiment is to determine the effects of a non-thrust manipulation procedure on muscle function, spinal mobility, and pain level on those experiencing low back pain (LBP) in a sample of individuals who identify English as their primary language. The rationale for this language criterion is provided in Section 9:F of this application. Muscle function will be measured via the muscle thickness of a deep spinal stabilizing muscle (multifidus, MF) while in both a resting state and during a maximum voluntary contraction (MVC). Spinal mobility will be measured as the active range of motion of both forward and backward trunk bending. Pain level will be a self-report measure recorded during rest and active range of motion.

Hypothesis 1: A non-thrust manipulation procedure will increase the thickness of the sacral multifidus both at rest and during a maximum voluntary contraction

Hypothesis 2: A non-thrust manipulation procedure will result in greater low back active range of motion.

Hypothesis 3: A non-thrust manipulation procedure will result in a reduction in the participant's self-reported pain levels both at rest and during active range of motion movements.

DETAILED DESCRIPTION:
The proposed study aims to determine if the impact of a newly-described manual procedure, that includes a non-thrust force applied to the low back region, has an impact on patient centered-outcomes. Rehabilitation Ultrasound Imaging (RUSI) will be used to determine MF muscle thickness (MT) at rest and during a maximum voluntary contraction (MVC) immediately following application of the manual procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are individuals with current complaint of low back pain, defined as pain that is present in the region from just below the rib cage to just below the buttocks.
2. Participants will be 18 years of age or older
3. Participants must be experiencing an episode of low back pain at the present time that is at any level on a Numerical Pain Rating Scale & Pain Diagram (NPRS) from 1-10
4. Participants must demonstrate the ability to maintain standing and prone postures for several minutes at a time and perform lumbar active range of motion in a standing position
5. Participants must report the presence of their low back pain during performance of active forward and/or backward bending in standing
6. Participants must demonstrate the ability to communicate in conversational English, that includes speaking, reading, and writing.

Exclusion Criteria:

1. Participants who are currently involved in litigation that is directly related to the participant's current episode of low back pain
2. Participants with known or suspected pregnancy
3. Participants with confirmed diagnosis of any of the following conditions:

   * Central nervous system disorder
   * Rheumatoid Arthritis
   * Spinal Fracture
   * Spondyloarthropathy (i.e., Ankylosing Spondylitis)
   * Tumor or infection of the spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Changes in Sacral Multifidus Muscle Thickness | Change from Pre to immediately Post Manipulation/Sham
  Rehabilitation Ultrasound Images of Sacral Multifidus muscle thickness at rest and during a maximal isometric contraction

SECONDARY OUTCOMES:
Changes in Lumbar Active Range of Motion | Change from Pre to immediately Post Manipulation/Sham
  Inclinometry of Lumbar Active Range of Motion in Standing
Changes in Low Back Pain | Change from Baseline to immediately Post Manipulation/Sham to 24-48 hours post session
  Visual Analogue Scale of Low Back Pain (0-10 scale with 0=least pain, 10=worst pain)
Changes in Oswestry Disability Questionnaire (0-100 scale, 0=no disability, 100=bed bound, exaggerating symptoms) | Change from Baseline to 24-48 hours post session
  Self-assessment disability paper survey
Changes in Fear-Avoidance Beliefs Questionnaire (0-96, 96=maximum fear-avoidance beliefs) | Change from Baseline to 24-48 hours post session
  Self-assessment disability paper survey
Changes in Global Rating of Change (-7 to +7 scale, -7=a very great deal worse, +7=a very great deal better) | Change from Baseline to 24-48 hours post session
  Self-assessment disability paper survey

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Cleland, PhD, Study Chair — Nova Southeastern University
Locations (1):
- Alvernia University, Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No